CLINICAL TRIAL: NCT06896058
Title: Effect of ınformatıon gıven to caregıvers of Stroke patıents wıth Percutaneous endoscopıc Gastrostomy on Care Burden and Self-care affaırs: a randomızed Controlled trıal
Brief Title: Effect of ınformatıon to caregıvers of Stroke patıents wıth Percutaneous endoscopıc Gastrostomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ceylan Kisial, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 26.10.2023-2903
Record Dates: First submitted 2024-11-29; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Progressing Stroke
Keywords: stroke patient with peg; care burden; self-care agency; information
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Experimental and control groups will be created
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Sham Comparator): The routine practices of the clinic (nutrition training is shown once by the service nurse) are applied to the relatives of the patients in the control group. No practices will be performed by the researcher. The relatives of the patients in both groups will be called by the researcher on the 15th and 30th days after discharge and the Burden Interview Scale (Appendix-2) and Self-Care Ability Scale (Appendix-3) will be applied. Thus, all relatives of the patients will be evaluated before and after the information. All evaluations and trainings will be performed by the same researcher to ensure standardization of the data.
  Interventions: Other: Written and verbal training given to caregivers
- Experimental group (Active Comparator): On the first day that the patients in the intervention group go to the palliative ward, the researcher will inform the relatives about care with a face-to-face education brochure. This information will take approximately 20 minutes. The researcher will call the relatives of the patients on the 15th and 30th days after discharge. In these calls, the necessary information will be repeated about the issues that the relatives need regarding care. These calls are estimated to take approximately 5 minutes. The researcher will call the relatives of the patients in both groups on the 15th and 30th days after discharge and apply the Burden Interview Scale (Appendix-2) and Self-Care Ability Scale (Appendix-3). In this way, all relatives of the patients will be evaluated before and after the information. All evaluations and trainings will be carried out by the same researcher to ensure standardization of the data.
  Interventions: Other: Written and verbal training given to caregivers

INTERVENTIONS:
Other: Written and verbal training given to caregivers — Education was provided with a brochure containing information on practices regarding care of stroke patients with PEG, prepared by the researcher in line with literature information.

SUMMARY:
Stroke is one of the serious neurological disorders that occur due to decreased blood flow to a certain part of the brain due to vascular injuries. Stroke ranks second in Europe among the causes of death in the world, fourth in the USA and second in Turkey. More than half of these patients who continue to live become partially or completely dependent on others for self-care and daily living activities. During this process, self-care is of critical importance in patients performing daily living activities and preventing complications. Self-care and needs of these patients are usually met by family members or relatives. The continuous care and needs of patients who are dependent or semi-dependent in self-care and daily living activities cause caregivers to have difficulty and experience burnout syndrome. This situation negatively affects caregivers physiologically, psychologically, socially and economically. The impact of all these negative situations on the caregiver and the difficulty they experience while providing care are defined as caregiver burden in the literature. If this burden causes the caregiver individual to have difficulty in performing their own daily living activities, it causes the caregiver's self-care ability to decrease or even be unable to perform them. As a result of the literature review, it was noticed that studies evaluating the difficulties experienced by caregivers and their self-care were generally conducted with caregivers who care for individuals with chronic diseases such as oncology and Alzheimer's. For this reason, determining the caregiver burden and providing regular support to caregivers, and providing planned training and counseling can help to suggest solutions to all these problems. Therefore, the aim of the study is to examine the effect of information provided to caregivers of stroke patients on the care burden and self-care ability.çalışmayı kabul etmeyen hastaların yakınları çalışmaya dahil edilmedi.

DETAILED DESCRIPTION:
Stroke is one of the serious neurological disorders that occur due to decreased blood flow to a certain part of the brain due to vascular injuries. Stroke ranks second in Europe among the causes of death in the world, fourth in the USA and second in Turkey. More than half of these patients who continue to live become partially or completely dependent on others for self-care and daily living activities. During this process, self-care is of critical importance in patients performing daily living activities and preventing complications. Self-care and needs of these patients are usually met by family members or relatives. The continuous care and needs of patients who are dependent or semi-dependent in self-care and daily living activities cause caregivers to have difficulty and experience burnout syndrome. This situation negatively affects caregivers physiologically, psychologically, socially and economically. The caregiver's being affected by all these negative situations and having difficulty while providing care is defined as caregiver burden in the literature. If this burden causes the caregiver individual to have difficulty in performing their own daily life activities, it causes the caregiver's self-care ability to decrease or even to be unable to perform them. At the same time, it shows that caregivers experience stress and burnout due to inadequacy in coping with patients' symptoms, unexpected needs arising during the care process, and this process causes changes in the caregivers' lives. Since most individuals have to continue their professional and social roles in addition to being caregivers, their areas of responsibility expand, their quality of life is negatively affected, and they may experience burnout due to changes in their free time and work-related activities. There are a limited number of outdated studies on family caregivers of stroke patients, and these studies reported that the care process has negative effects on the health and well-being of caregivers. Due to the sudden onset of disability and the chronic nature of recovery from stroke, caring for a stroke patient has been found to have a negative impact on the physical, mental, and psychological health of caregivers. As a result of the literature review, it was noticed that studies evaluating the difficulties experienced by caregivers and their self-care were generally conducted with caregivers who care for individuals with chronic diseases such as oncology and Alzheimer's. For this reason, determining the caregiver burden and providing regular support to caregivers, and providing planned training and counseling can help to suggest solutions to all these problems. Therefore, the aim of the study is to examine the effect of information provided to caregivers of stroke patients on the care burden and self-care ability.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older, conscious, person-time and place oriented,
* No psychiatric problems, no hearing-speech or visual impairments,
* Can speak Turkish,
* Patient relatives who accompany the patient in the hospital environment and will continue to provide care at home and who accept the research were included.

Exclusion Criteria:

* Relatives of patients who could not be contacted,
* Resulted in death,
* Did not accept the study were not included in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Burden of Care Scale (Burden Interview) | 1 year
  The scale provides a minimum (0) and maximum (88) score. As the score increases, the difficulty experienced by the patient's relative in his/her life increases.
Determining the caregiver burden and providing regular support to caregivers, planned training and counseling can help find solutions to all these problems. | 1 year
  The Caregiver Diagnosis Form, Caregiver Burden Scale and Self-Care Ability Scale, as well as written training materials and brochures, were used.
  As the score increases, the difficulty experienced by the patient's relative in his/her life increases.